CLINICAL TRIAL: NCT06501911
Title: Phase I Dose Escalation Study on Bicalutamide, an Androgen Receptor Antagonist, as a Radiosensitizer Combining With Brain Re-irradiation to Treat Recurrent/Progressive Glioblastoma/High Grade Glioma
Brief Title: A Study of Bicalutamide With Brain Re-irradiation to Treat Recurrent/Progressive High Grade Glioma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI leaving institution.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0608-24-FB
Record Dates: First submitted 2024-07-05; First posted 2024-07-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Glioblastoma; Recurrent High-grade Glioma
Keywords: Progressive high grade glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — bicalutamide; Radiotherapy, Intensity-Modulated; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bicalutamide with brain re-irradiation (Experimental): Participants will take oral bicalutamide daily for six (6) months at a starting dose of 150 mg daily. Participants will be enrolled in cohorts of six (6) participants. The dose will be incrementally adjusted based on dose limiting toxicities seen in the previously enrolled cohort until the Maximum Tolerated Dose (MTD) is reached. The MTD is defined as the dose level below the dose at which at least two (2) of six (6) participants experienced a dose limiting toxicity.
  Participants will also receive 10 fractions of brain re-irradiation beginning one week after the start of bicalutamide treatment.
  Interventions: Drug: Bicalutamide; Radiation: Intensity-modulated radiation therapy (IMRT)

INTERVENTIONS:
Drug: Bicalutamide — Participants will receive daily oral bicalutamide for six (6) months. The dose will be determined by the cohort to which the participant is enrolled as well as the toxicities experienced by previously enrolled cohorts.
  Other Names: Casodex
Radiation: Intensity-modulated radiation therapy (IMRT) — Participants will receive 35 Gy delivered in 10 fractions, administered once daily on weekdays.
  Other Names: Three-Dimensional Conformal Radiation Therapy (3D-CRT)

SUMMARY:
The goal of this study is to learn about a type of brain cancer called high-grade glioma. This study is for people who have previously received treatment for brain cancer, but the cancer has come back or gotten worse after treatment. The main question this study aims to answer is: is it safe for participants to take bicalutamide while receiving brain radiation treatment?

Participants will:

* Take bicalutamide every day for 6 months
* Receive radiation treatment to the brain
* Keep a diary of the when they take the bicalutamide and any side effects experienced
* Visit the clinic once every 8 weeks for checkups and tests

DETAILED DESCRIPTION:
Participants will be enrolled according to a standard cohort 3+3 dose-escalation/de-escalation study design at a starting dose of 150 mg of bicalutamide. Up to six (6) subjects will be enrolled to a given dose level until the Maximum Tolerated Dose (MTD) is reached, or until a maximum dose of 600 mg is reached. The MTD is defined as the dose below which two (2) or more of six (6) subjects experience a dose limiting toxicity (DLT). If the starting dose exceeds the MTD, the dose will be decreased until a minimum dose of 25 mg is reached.

Primary Objective:

1. To evaluate the safety when combining partial brain re-irradiation with bicalutamide. Side effects of the study drug combined with radiation therapy (RT) will be assessed per CTCAE 5.0.

Secondary Objectives:

1. To estimate the rate of objective response rate (ORR) in subjects with treatment. Response Assessment in Neuro-Oncology (RANO) criteria will be used to estimate ORR.
2. To estimate the 6-month progression-free survival rate.
3. To evaluate the impact of combining bicalutamide with brain re-irradiation on quality of survival, as measured by changes to scores on the Montreal Cognitive Assessment (MoCA) and Karnofsky performance status.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of relapsed/refractory high-grade glioma (HGG) including glioblastoma or variants (gliosarcoma, giant cell glioblastoma etc), World Health Organization (WHO) grade IV, or anaplastic astrocytoma, or anaplastic oligodendroglioma, WHO grade III. Participants will be eligible if the original histology was lower-grade glioma and a subsequent diagnosis of HGG (secondary HGG) is made.
* Participants who did not have surgery for their HGG within 5 weeks prior to enrollment must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced magnetic resonance imaging (MRI) scan (or CT scan for participants with non-compatible devices). Imaging completed prior to enrollment will be acceptable for eligibility purposes if completed within 4 weeks prior to enrollment. If imaging was not completed within 4 weeks prior to enrollment then imaging must be completed within 14 days after enrollment and prior to the start of RT.

Participants unable to undergo magnetic resonance (MR) imaging because of non-compatible devices can be enrolled provided CT scans are obtained and are of sufficient quality. Participants without non-compatible devices may not use CT scans performed to meet this requirement.

* Participants must have passed an interval of 6 months or greater between completion of prior radiotherapy and enrollment. If participants have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

  * New areas of tumor outside the original radiotherapy fields as determined by the investigator
  * Histologic confirmation of tumor through biopsy or resection
  * Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of previous radiotherapy and registration
* Prior history of standard dose central nervous system (CNS) radiation of 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent or lower doses.
* Participants must have recovered from the toxic effects of prior chemotherapy, and there must be a minimum time of 14 days prior to enrollment from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:

  * 14 days from administration of vincristine
  * 42 days from administration of nitrosoureas
  * 21 days from administration of procarbazine
* Participants having undergone recent resection of their glioblastoma (within 5 weeks prior to enrollment) must have recovered from the effects of surgery. For CNS related core or needle biopsies, a minimum of 7 days must have elapsed prior to enrollment.

Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study.

* History/physical examination, including neurologic examination, within 14 days prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) ≤ 2 within 14 days prior to enrollment
* Age ≥ 19 (Age of majority in Nebraska)
* Complete blood count (CBC)/differential obtained within 14 days of enrollment, with adequate bone marrow function. Adequate bone marrow reserve as follows:

  o Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 Platelets ≥ 75,000 cells/mm3 Hemoglobin ≥ 9.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable.) Note: If a CBC w/differential was not obtained prior to enrollment it must be completed within 14 days of enrollment and prior to the start of bicalutamide.
* Acceptable liver (total bilirubin < 2.0 mg/dL, and glutamic-oxaloacetic transaminase (SGOT) or Aspartate Transferase (AST) < 2.5 times the upper limit of normal) and renal function [serum creatinine < 1.8 mg/dL and calculated creatinine clearance > 30 ml/min (Cockroft-Gault)] within 14 days of enrollment. Note: If labs were not completed prior to enrollment they must be completed within 14 days of enrollment and prior to the start of bicalutamide.
* Urine protein: creatinine (UPC) ratio < 1.0 OR urine dipstick for proteinuria ≤ 2+ completed within 14 days of enrollment. If not completed prior to enrollment it must be completed within 14 days and prior to the start of bicalutamide. Note: Participants discovered to have > 2+ proteinuria on dipstick urinalysis at baseline must have a UPC ratio done that is <1.0 to be eligible. If the UPC ratio is ≥ 1.0 then the Participants will undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible. If a 24-hour urine collection is necessary it must be completed within 14 days of enrollment and prior to the start of bicalutamide. Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. UPC ratio is calculated using one of the following formulas:

  * [urine protein]/[urine creatinine]: if both protein and creatinine are reported in mg/dL
  * [(urine protein) x0.088]/[urine creatinine]: if urine creatinine is reported in mmol/L
* Participants must not be pregnant (positive pregnancy test) or breast feeding; pregnancy test must be done within 7 days of enrollment and prior to the start of RT. Effective contraception (men and women), i.e., effective physical barrier methods, must be used in subjects of child-bearing potential while on study treatment and for 6 months after. Oral contraceptives are not allowed as a form of contraception due to potential interference of testosterone levels.
* Participants on full-dose anticoagulants [e.g., warfarin or low molecular weight heparin (LMW) heparin] must meet both of the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * In-range international normalised ratio (INR) (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, within 14 days of enrollment and prior to the start of bicalutamide
* Participants must be able to provide study-specific informed consent prior to study entry.

Exclusion Criteria:

* Infratentorial, or diffuse leptomeningeal evidence of recurrent disease. If focal leptomeningeal disease (per treating physician's determination of being "focal"), participants can be considered eligible.
* Ongoing therapy with any androgen deprivation therapy (ADT) such as leuprolide acetate, degarelix, bicalutamide, flutamide, enzalutamide, apalutamide, abiraterone acetate, darolutamide or others per principal investigator's determination. If ADT has been stopped prior to the enrollment, at least 6 months of ADT-free time is required for eligibility.
* Prior allergic reaction to the drug bicalutamide 3.2.4 Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (for example, carcinoma in situ of the breast, oral cavity, prostate, or cervix are all permissible).
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration.
  * Congestive heart failure (NYHA functional capacity class II or greater).
  * Transmural myocardial infarction within the last 6 months prior to registration.
  * History of stroke or transient ischemic attack within 6 months prior to registration.
  * Ongoing arrhythmias of Grade >2 [CTCAE, version 5.0]; Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
  * Thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism) in the past 6 months.
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
  * Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed. 3.2.6 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
* Known Acquired Immune Deficiency Syndrome (AIDS) diagnosis based upon current Centers for Disease Control (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude participants with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
* Immuno-compromised participants with transplant in history are excluded.
* Uncontrolled seizures or controlled seizure in the past 3 months but requires more than levetiracetam 500mg orally twice a day, i.e., with higher dose of levetiracetam or additional antiepileptics (excluding steroids).
* Any prior history of hypertensive crisis or hypertensive encephalopathy. 3.2.12 History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to enrollment 3.2.13 Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse.
* Participants who are on testosterone supplement due to medical reasons that cannot be safely discontinued.
* Participants who are on temozolomide treatment and have no plan to stop temozolomide prior to consent or who will be offered temozolomide concurrently with re-RT. Subjects on bevacizumab whose bevacizumab cannot be stopped are not eligible and bevacizumab is not allowed for concurrent use with bicalutamide and re-RT but is allowed after at least two weeks (washout time) after discontinuation of re-RT and bicalutamide.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) in participants receiving study treatment (combining partial brain re-irradiation with bicalutamide) | Up to 26 months
  The incidence of adverse events (AEs) will be described for each dose level cohort as well as the two highest dose levels combined. Toxicities will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicities will be graded on a scale ranging from 1 to 5, with higher numbers indicating a higher severity grade.
The incidence of serious adverse events (SAEs) in participants receiving study treatment (combining partial brain re-irradiation with bicalutamide) | Up to 26 months
  The incidence of serious adverse events (SAEs) will be described for each dose level cohort as well as the two highest dose levels combined. Toxicities will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicities will be graded on a scale ranging from 1 to 5, with higher numbers indicating a higher severity grade.

SECONDARY OUTCOMES:
Rate of objective response (ORR) in participants receiving treatment | Up to 44 months
  The rate of objective response (ORR) in subjects receiving treatment will be assessed using Response Assessment in Neuro-Oncology (RANO) Criteria. MRI and clinical features are used to classify response as one of four categories that range from complete response to disease progression.
Six-month Progression-free Survival Rate | Up to 26 months
  Progression-free survival (PFS) will be estimated using the Kaplan-Meier method which estimates event probability occurring at a specific time point among subject who have not already experienced that event. PFS is defined as the time from the date of consent to disease progression or death.
The impact of study treatment on quality of survival (Montreal Cognitive Assessment) | Up to 44 months
  To evaluate the impact of combining bicalutamide with brain re-irradiation on the quality of survival, score changes on the Montreal Cognitive Assessment (MoCA) will be measured at protocol-specified time points throughout the study. Maximum score on the assessment is 30 (scores of 30 to 26 indicate no impairment, 25 to 18 mild cognitive impairment, 17 to 10 moderate cognitive impairment, less than 10 severe cognitive impairment.
The impact of study treatment on quality of survival (Karnofsky Performance Scale) | Up to 44 months
  To evaluate the impact of combining bicalutamide with brain re-irradiation on the quality of survival, scores changes on the Karnofsky Performance Scale will be measured. This scale ranges from 0 to 100: 100 indicates normal health and survival decreases with decreasing scores.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Zhang, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No